CLINICAL TRIAL: NCT04343313
Title: Evaluation of the Safety and Performance of the Half Moon Transcatheter Mitral Valve Repair System in High Risk Patients With Severe, Symptomatic Mitral Regurgitation
Brief Title: The Half Moon Transcatheter Mitral Valve Repair (TMVr) Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Half Moon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0001
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Half Moon TMVr System (Experimental): The Half Moon Transcatheter Mitral Valve Repair (TMVr) System is designed for transfemoral access and transseptal delivery of a self-expanding implant that restores competency in a regurgitant mitral valve.
  Interventions: Device: Half Moon TMVr System

INTERVENTIONS:
Device: Half Moon TMVr System — The Half Moon Transcatheter Mitral Valve Repair (TMVr) System is designed for transfemoral access and transseptal delivery of a self-expanding implant that restores competency in a regurgitant mitral valve.

SUMMARY:
The study is a prospective, multi-center, single-arm, non-randomized, Early Feasibility Study (EFS) to evaluate the safety and performance of the Half Moon TMVr System in patients with severe, symptomatic mitral regurgitation, who are at high risk for conventional mitral valve surgery.

ELIGIBILITY:
Key Inclusion Criteria:

1. Moderately severe or severe mitral regurgitation (MR Grade ≥ 3+)
2. Symptomatic mitral regurgitation (NYHA Class II-IV), despite guideline-directed medical therapy (GDMT) determined by the local multidisciplinary heart team
3. Deemed, by the local multidisciplinary heart team, to be at high risk for mitral valve surgery and not appropriate for commercially approved transcatheter mitral valve therapies
4. Age ≥ 21
5. Native mitral valve geometry and size compatible with the Half Moon TMVr implant
6. Anatomy suitable for transfemoral transseptal access with the Half Moon TMVr System
7. Willing to sign Informed Consent for participation in the study and return for all required post-procedure follow-up visits

Key Exclusion Criteria:

1. Prior transseptal intervention with occlusion device currently implanted
2. Implanted with venous stents (iliac and femoral) including inferior vena cava (IVC) filter or congenital abnormalities of the IVC that would preclude ability for transfemoral access with the delivery system
3. Evidence of intracardiac, inferior vena cava, or femoral venous mass, thrombus, or vegetation
4. Prohibitive mitral annular or leaflet calcification
5. Diseased mitral anterior leaflet such as flail or prolapse
6. Left ventricular ejection fraction (LVEF) < 25%, or LVEF 25-30% in the presence of left ventricular end diastolic volume index (LVEDVi) >120mL/m2 as measured by resting echocardiogram within 30 days of the Index Procedure
7. Left ventricular end diastolic diameter (LVEDD) > 75mm
8. Pulmonary hypertension with resting pulmonary artery systolic pressures ≥ 2/3 systemic systolic pressure
9. Right-sided congestive heart failure with echocardiographic evidence of severe right ventricular dysfunction
10. Severe tricuspid regurgitation
11. Prior mitral valve surgery or endovascular procedure, or need for other valve surgery/procedure
12. Any endovascular therapeutic interventional or surgical procedure performed within 30 days prior to enrollment
13. Prior stroke, TIA, or myocardial infarction within 90 days
14. Need for coronary revascularization
15. Severe symptomatic carotid artery stenosis
16. Severe Chronic Obstructive Pulmonary Disease (COPD) demonstrated by Forced Expiratory Volume (FEV1) < 750cc
17. Need for emergent surgery
18. Endocarditis within 6 months
19. Subject is unwilling or unable to adhere to the protocol recommended anticoagulation treatment
20. GI bleeding within 6 months
21. History of bleeding diathesis or coagulopathy or patient will refuse blood transfusion
22. Hemodynamic instability requiring dependency on either inotropic agents or mechanical circulatory support
23. Platelet count of <75,000 cells/mm3
24. Renal insufficiency (Creatinine > 2.5 mg/dL)
25. Active infections requiring current antibiotic therapy (if temporary illness, patients may enroll 2 weeks after discontinuation of antibiotics)
26. Contraindication to transesophageal echocardiography (TEE)
27. Known hypersensitivity or contraindication to study or procedure medications/contrast which cannot be adequately managed medically
28. Pregnant, nursing or planning to be pregnant. (Female participants of childbearing potential must have a negative pregnancy test prior to enrollment)
29. Currently participating in an investigational drug or another device study that has not yet reached its primary endpoint

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 30 Days
  Evaluation of the nature, severity and frequency of complications associated with the delivery and/or implantation of the device

SECONDARY OUTCOMES:
Device Placement | 30 Days (+ annually through 5 years)
  Assessment of the ability to accurately deliver and place the implant within the native anatomy
Device Performance | 30 Days (+ annually through 5 years)
  The degree of improvement of MR grade
Symptom Improvement | 30 Days (+ annually through 5 years)
  The degree of improvement of MR symptoms
Device Durability | 30 Days (+ annually through 5 years)
  The durability of TMVr function

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Heart & Vascular Institute, Harrisburg, Pennsylvania